CLINICAL TRIAL: NCT02219841
Title: Impact of Life-Style Modification On Ablation Outcome in Atrial Fibrillation
Acronym: ISOLATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: TCAI_ISOLATE
Record Dates: First submitted 2014-07-31; First posted 2014-08-19 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation; Obesity
Keywords: Obesity, low-calorie diet, exercise, atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Motor Activity | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No intervention group: Receive general life-style advice and information on heart healthy diet Undergo catheter ablation for AFib
  Interventions: Procedure: radiofrequency catheter ablation
- Life-style intervention: patients will receive personilized low-calorie diet menu and undergo supervised exercise in the cardiac rehabilitation facility for 3 months before ablation with an aim of loosing >10% of body weight. They will continue diet and exercise for 1 year following ablation procedure Will receive catheter ablation for AFib
  Interventions: Procedure: radiofrequency catheter ablation

INTERVENTIONS:
Procedure: radiofrequency catheter ablation
  Other Names: RFCA

SUMMARY:
This prospective randomized pilot study aims to evaluate the impact of aggressive life style modification in terms of calorie-controlled diet and supervised exercise on outcome of catheter ablation in overweight and obese patients with atrial fibrillation.

Hypothesis: Weight loss and management by adoption of strict diet and exercise regimen improves the chances of freedom from recurrence following catheter ablation.

DETAILED DESCRIPTION:
Objective: To examine the impact of a planned life-style modification program including calorie-controlled diet and supervised exercise before and after the AF ablation on quality of life (QoL) and long-term arrhythmia recurrence in overweight and obese patients with atrial fibrillation.

Endpoints:

Primary: AF recurrence following index ablation procedure It will be assessed at 3, 6 and 12 months after the procedure by event recorders, 12-lead ECG and Holter monitoring Any episode of AF/AFL/AT > 30 sec will be considered as a recurrence. Episodes that occur during the first 3 months after the procedure (blanking period) will not be considered as recurrence.

Secondary:

1. Change in QoL It will be evaluated by a validated AF specific questionnaire (AFEQT) at baseline and 6 and 12 months post-procedure
2. Change in AF symptom severity. This will be measured by AF symptom severity and burden questionnaire at baseline and 6 and 12 months post-procedure

DIET:

Participants in the intervention group will receive individual counseling sessions with an experienced dietitian, who will prepare personalized diet plan based on their comorbidities and preferences.

To accomplish weight loss, the diet menu will be planned to reduce daily food intake by ≥ 500 calories depending on their baseline body weight.

Patients enrolled in the control group will be provided advice on heart-healthy diet and active life style.

EXERCISE:

Supervised and monitored exercise will be conducted in St. David's Cardiac Rehabilitation for 3 months starting before or 7-10 days after the ablation.

After ablation, patients will continue individualized home-exercise program for 1 year.

QoL Survey:

The AF Effect on Quality of Life survey (AFEQT) questionnaire will be used at baseline and 6 and 12 months post procedure.

Symptom Severity Survey:

This will be measured by AF symptom severity and burden questionnaire at baseline and 6 and 12 months post-procedure

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 18 years
2. AF patient undergoing first catheter ablation, at least 3 months after the enrollment
3. BMI: ≥ 26-40
4. Willing to be compliant with the weight-reduction program
5. Willing to provide informed, written consent

Exclusion Criteria:

1. Chronic obstructive lung disease (COPD)
2. Participation in another weight loss program in < 3 months
3. Musculoskeletal conditions limiting exercise capacity
4. Insulin-dependent diabetes
5. Severe valvular heart disease or cardiomyopathy
6. Heavy drinking (>14 standard drinks/week for men and >7/ week for women)
7. Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 consecutive AF patients with BMI 26-40, will be enrolled in this pilot study and randomized to 2 groups in a 1:1 design (25 per group).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 1 year post-ablation
  Arrhythmia recurrence will be monitored at 3-month intervals with Holter monitor, event recorder, cardiology evaluation and ECG. Recurrence is defined as any episode of AF/ atrial flutter/ atrial tachycardia of >30 seconds duration with or without anti-arrhythmic drugs, occurring after 3 months of blanking period following catheter ablation

SECONDARY OUTCOMES:
Quality of Life | 1 year
  The AF Effect on Quality of Life survey (AFEQT questionnaire will be used at baseline and 6 and 12 months post procedure. It is a validated self-administered questionnaire of 20 questions for AF patients that evaluates health-related QoL across 3 domains; symptoms, daily activity and treatment concerns

OTHER OUTCOMES:
Weight loss | 1 year
  Weight loss following calorie-controlled diet and monitored exercise for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Mitra Mohanty, MD, Principal Investigator — Texas Cardiac Arrhythmia Institiute
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. david's Medical Center, Austin, Texas, United States